CLINICAL TRIAL: NCT05316909
Title: Effect of a Newborn Simulator's Fidelity on Nursing Students' Level of Engagement in a Clinical Lactation Encounter
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Alternate study completed
Sponsor: LiquidGoldConcept (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 21-003
Record Dates: First submitted 2022-03-18; First posted 2022-04-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Breastfeeding; Education, Nursing
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: Educational intervention with newborn simulators of varying fidelity
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are unaware of their intervention assignment (order of dolls).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baby doll with remote controlled jaw (Experimental): In this arm, standardized patients will use the Newborn Oral Assessment and Latch Simulator (NORALSim) to demonstrate and teach newborn positioning and attachment in the simulation.
  Interventions: Other: Breastfeeding Simulation
- Standard care/doll (Active Comparator): In this arm, standardized patients will use a cloth doll/standard treatment to demonstrate and teach newborn positioning and attachment in the breastfeeding skills workshop.
  Interventions: Other: Breastfeeding Simulation

INTERVENTIONS:
Other: Breastfeeding Simulation — In Period 1, one group will begin a simulated session with the NORALSim and the second group will begin with either the Mother's Own Milk Lactessa or Laerdal NeoNatalie, depending on the study date. Baseline level of breastfeeding experience and clinical lactation skills self-efficacy will be collected. Nursing students will teach a mock patient wearing the LSM and holding a newborn simulator how to position and attach the newborn at the breast and identify effective breastfeeding by differentiating between suckling patterns. In Period 2, each group will crossover to complete the same session with a different newborn simulator. After Period 1, each group will debrief to discuss their performance and engagement and use a Qualtrics survey (6-point Likert scale) to rate satisfaction, engagement, simulator fidelity, and self-efficacy. The same quantitative and qualitative data collection protocol will follow Period 2.

SUMMARY:
Nursing students (N=32) will be randomized to begin period 1 in either a high-fidelity or low-fidelity simulated experience with a mock patient wearing a breast model and holding a newborn simulator and then cross over in period 2 to the opposite arm. Data on student satisfaction, engagement, self-efficacy, and performance and simulator fidelity will be collected via Qualtrics surveys (defined, 6-point Likert scale), written and oral reflection, audio-video recordings of clinical lactation encounter, and clinical lactation skills checklists and global performance ratings.

Nursing students in the accelerated master's program will be recruited while completing their required simulation coursework. A random number generator will be used to randomly assign students to a treatment arm. Investigators will require at least 8 students per arm (power 80%, alpha 5%). Investigators will recruit 32 students for two study dates to compare the high-fidelity LiquidGoldConcept products to two competitor products.

The Johns Hopkins School of Nursing and Simulation Center will be the only sites where human subjects research will be performed. The collaborating investigators (Drs. Debbie Busch, Joanne Silbert-Flagg, and Nancy Sullivan) have expertise in clinical lactation education and simulation. With the collaborating investigators LiquidGoldConcept has already completed pilot studies to establish the feasibility of our approach and validate the survey instruments.

DETAILED DESCRIPTION:
This is a randomized cluster design intervention. Assuming an enrollment ratio of 1, alpha of 0.05, beta of 0.2, investigators will recruit at least 8 students per arm with 16 students in the NORALSim arm and 16 students low-fidelity newborn simulator arm. A random number generator will be used to assign students to a study ID number (1-32). Students will be randomly assigned to a group of four a priori by assigning each student a number between 1 and 4. Three mock patients will be randomized a priori to minimize the confounding effect of a mock patient's acting abilities. Approximate start times are as follows: Groups 1 and 2 will begin at 8:30AM, Groups 3 and 4 will begin at 10AM, Groups 5 and 6 will begin at 1pm, and groups 7 and 8 will begin at 2:30pm. Investigators will alternate the order of the low-fidelity simulators (Lactessa or NeoNatalie) and randomize that order a priori such that 8 students (2 groups) will interact with the Lactessa and another 8 students (2 groups) will interact with Neonatalie.

In Period 1, one group will begin a simulated session with the NORALSim and the second group will begin with either the Mother's Own Milk Lactessa or Laerdal NeoNatalie, depending on the study date. Baseline level of breastfeeding experience and clinical lactation skills self-efficacy will be collected. Nursing students will teach a mock patient wearing the LSM and holding a newborn simulator how to position and attach the newborn at the breast and identify effective breastfeeding by differentiating between suckling patterns. In Period 2, each group will crossover to complete the same session with a different newborn simulator. After Period 1, each group will debrief to discuss their performance and engagement and use a Qualtrics survey (6-point Likert scale) to rate satisfaction, engagement, simulator fidelity, and self-efficacy. The same quantitative and qualitative data collection protocol will follow Period 2. All study activities will be audio-video recorded. JHU investigators will view the recorded encounters and assign a performance score using a skills checklist and global performance rating scale. Within a month, students will view their clinical encounters recording and complete a self-reflection to describe moments of engagement or disengagement. Students will also report any breastfeeding experience obtained since the intervention, score their performance, and complete the self-efficacy survey.

ELIGIBILITY:
Inclusion Criteria:

* Student enrolled at Johns Hopkins University School of Nursing

Exclusion Criteria:

* Younger than 18
* Not able to complete study activities

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Level of Engagement | Immediately after intervention
  The primary outcome is the level of engagement. A level of engagement score will be calculated from one qualitative and three quantitative criteria: 1) student self-reported perception of engagement during debriefing and self-reflection (qualitative), 2) time to task completion in both periods (quantitative, defined 6-point Likert scale in Qualtrics survey), 3) engagement survey score after both periods (quantitative, defined 6-point Likert scale in Qualtrics survey), and 4) global performance ratings by JHU faculty and students (quantitative, 4-item, 8-points possible).
Level of Engagement | One Month
  The primary outcome is the level of engagement. A level of engagement score will be calculated from one qualitative and three quantitative criteria: 1) student self-reported perception of engagement during debriefing and self-reflection (qualitative), 2) time to task completion in both periods (quantitative, defined 6-point Likert scale in Qualtrics survey), 3) engagement survey score after both periods (quantitative, defined 6-point Likert scale in Qualtrics survey), and 4) global performance ratings by JHU faculty and students (quantitative, 4-item, 8-points possible).

SECONDARY OUTCOMES:
Satisfaction with the simulation experience | Immediately after intervention
  Students' satisfaction after both periods (quantitative, defined 6-point Likert scale in Qualtrics survey)
Self-Efficacy in clinical lactation/breastfeeding skills | Immediately after intervention
  Student self-efficacy in clinical lactation skills (quantitative, defined 6-point Likert scale in Qualtrics survey).
Student performance of breastfeeding skills | Immediately after intervention
  Student performance (in both periods) using clinical lactation skills checklist and global performance rating

CONTACTS AND LOCATIONS:
Locations (1):
- LiquidGoldConcept, Ypsilanti, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
Researchers do not plan to share IPD with other researchers.